CLINICAL TRIAL: NCT01735929
Title: Evaluating the Combined Skin Tightening Benefit of Non-Invasive Ultrasound Treatment and Neck Liposuction
Brief Title: Combination of Ultrasound Treatment and Neck Liposuction for Skin Tightening
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology- Head and Neck Surgery and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU68167
Record Dates: First submitted 2012-11-05; First posted 2012-11-28 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neck Liposuction and Ultrasound Treatment (Experimental): Subject will receive neck liposuction and ultrasound treatment.
  Interventions: Procedure: Neck Liposuction and Ultrasound Treatment
- Sham (Sham Comparator): Subject will receive sham treatment
  Interventions: Procedure: Sham Treatment

INTERVENTIONS:
Procedure: Neck Liposuction and Ultrasound Treatment
  Arms: Neck Liposuction and Ultrasound Treatment
Procedure: Sham Treatment
  Arms: Sham

SUMMARY:
The purpose of this study is to find out the effectiveness of ultrasound treatment and liposuction combined on skin tightening around the neck.

ELIGIBILITY:
Inclusion Criteria:

* Women 35-60 years old
* Exhibit mild to moderate neck skin laxity on clinical examination
* No other serious health problems, including psychiatric illness.

Exclusion Criteria:

* Prior neck surgery or face lift.
* Bleeding disorders or coagulopathy.
* Botulinum toxin or filler injections to neck area within past 6 months.
* Severe neck skin laxity or sagging
* Other serious medical conditions that in the opinion of the surgeon could compromise safety

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in photo ratings at 8 weeks. | Baseline and 8 weeks
  Two blinded raters will compare baseline and 8 week photos of subjects that received the combined treatments or the sham treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University